Title: Pilot Study to Evaluate the Anti-Tumor Effect of Durvalumab (Medi4736) in Patients With Squamous Cell Carcinoma of the Head and Neck (SCCHN), Human Papilloma Virus (HPV) Positive Versus Negative, When Treated Before Surgery

NCT02827838

Date: 6/28/21



Section of Hematology and Oncology

## PILOT STUDY TO EVALUATE THE ANTI-TUMOR EFFECT OF DURVALUMAB IN PATIENTS WITH SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK (SCCHN), HUMAN PAPILLOMA VIRUS (HPV) POSITIVE VERSUS NEGATIVE, WHEN TREATED BEFORE SURGERY

Informed Consent Form to Participate in Research Mercedes Porosnicu, MD, Principal Investigator

#### INTRODUCTION

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you have cancer of the head and neck.

This consent form gives you important information about this study to help you decide if you want to participate. It describes the purpose of this study, the study procedures, the possible risks, and provides information about your rights as a study participant.

Please take the time to read this information carefully. You should talk to the study doctor and his/her study staff about this study and ask to explain any words or information contained in this informed consent document that you do not understand and ask any questions you have. You can also discuss this study with other people such as your family or personal doctor. Please take your time in making your decision as to whether or not you wish to participate. If you decide to participate in this study, you will be asked to sign and date this form. You will receive a copy of the signed form.

If you have a different personal doctor, the study doctor will ask if he/she can tell your personal doctor about your participation in this study.

Your participation in this study is voluntary. You are free to say yes or no. If you do not want to participate, your regular medical care and legal rights will not be affected. Even if you join this study, you may stop at any time.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by US Law.

## WHY IS THIS STUDY BEING DONE?

You have been asked to take part in this study because you have a type of head and neck cancer which is called squamous cell carcinoma of the head and neck (SCCHN). The standard treatment for your condition is surgery. As you have already been informed, the date for your surgical treatment has been established and there is a waiting period before this can be performed. The purpose of this research study is to determine whether during this period of time, giving you an antibody in the form of a medication called Durvalumab (study drug) can hold your tumor from growing and to examine the effect of this study drug against your cancer. Durvalumab is approved for the treatment of locally advanced or metastatic urothelial cancers and for patients with stage III non-small cell lung cancer. Antibodies are proteins produced by



the defense system of the body (immune system) that have been made in the laboratory. This treatment helps increase the activity of the immune system that in many cases is decreased by the cancer. When the immune system is more active, it has a better chance to fight the cancer in your body, trying to limit the spread of the cancer. This medication is considered experimental for the treatment of SCCHN as it has not been yet approved by FDA.

This study has three goals. One goal is to measure how effective this treatment is to stop the growth of your tumor when given before your surgery. Another goal is to help find biologic molecules in the tumor or saliva or blood that prove to be good indicators of how efficient this medication is against your cancer. Using samples of blood and saliva collected before and after treatment as well as a small piece of tumor collected by biopsy before treatment with Durvalumab, and a piece of your tumor removed during the surgical treatment, we plan to make special analyses in the lab in order to find changes that can be used in the future to predict response to the Durvalumab medication. The third goal is to check if this medication is more or less effective in patients who have tumors positive or negative for a virus called Human Papilloma Virus (briefly HPV) that is present in many cancers of the head and neck.

## HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

20 people will take part in this study. 10 patients will have the tumor positive for the Human Papilloma Virus (HPV) and 10 patients will have the tumors negative for HPV.

## WHAT IS INVOLVED IN THE STUDY?

If you take part in this study, you will

- Receive Durvalumab twice before your scheduled surgery with 14 days between the two doses. If the time to your surgery is longer than 30 days, a third dose of treatment will be scheduled.
- Have the following tests and procedures during the Screening Visit (within 28 days prior to first drug administration):
  - o Demographic information, history of tobacco and alcohol use, medical history
  - o Physical exam, performance status assessment, vital signs, height, weight, EKG, current medications
  - Tumor biopsy
  - o Imaging by CT scan or MRI, PET scan
  - o Blood sample collection about two tablespoons of blood
  - Saliva sample collection: 5 ml of saliva will be collected by drooling into a large diameter tube.
  - o HPV test done in the tumor tissue
  - o Pregnancy test for women of childbearing potential
  - o As part of this study, you will be tested for HIV (human immunodeficiency virus, which is the virus that causes the acquired immunodeficiency syndrome [AIDS]); Hepatitis A, B, and C. You will be told of the results of the testing, and counseled as to the meaning of the results, whether they are positive or negative. If the test indicates that you are infected with one of these diseases, you will receive additional counseling about the significance of your care and possible risks to other people. We are required by law to report all positive results to the North Carolina State Board of Health. The test results will be released only as permitted by applicable law. If you do not want to be tested for these diseases, you should



not agree to participate in this study.

- Have the following tests and procedures during the First Drug Administration Visit (Week 1 of the study):
  - Receive durvalumab through a vein (peripheral or central line) administered over
     60 minutes
  - o Physical exam, performance status assessment, vital signs, height, weight, EKG, current medications
  - o Blood sample collection
  - Saliva sample collection
- Have the following tests and procedures during the Follow-up Visit 1 (Week 2 of the study):
  - Physical exam, performance status assessment, vital signs, height, weight, current medications
  - Blood sample collection
  - o Saliva sample collection
- Have the following tests and procedures during the Second Drug Administration Visit (Week 3 of the study):
  - Receive durvalumab through a vein (peripheral or central line) administered of 60 minutes
  - Physical exam, performance status assessment, vital signs, height, weight, current medications
  - Blood sample collection
  - o Saliva sample collection
- Have the following tests and procedures during the Follow-up Visit 2 (Week 4 of the study):
  - Physical exam, performance status assessment, vital signs, height, weight, current medications
  - Blood sample collection
  - o Saliva sample collection
- Have the following tests and procedures during the Pre-Surgery Visit (1-2 days before surgery):
  - Physical exam, performance status assessment, vital signs, height, weight, EKG, current medications
  - Blood sample collection
  - Saliva sample collection

Version: 07/11/19

o Imaging by CT scan or MRI, PET scan

Blood and saliva sample collection will be done in a similar fashion at each visit. You will have approximately 2 tablespoons – 35 ml of blood withdrawn from a vein with each visit. The total amount of blood withdrawn during the study will be approximately 10 tablespoons – 165 ml (6 ounces). It could be 4 tablespoons more in case the time window to your surgery is longer than 30 days.

# Collection, Storage and Use of Biological Tissue

You will then have surgical treatment as scheduled by your Ear, Nose and Throat (ENT)



surgeon. At the time of surgery, your tumor will be removed and carefully measured and evaluated by our Department of Pathology and all tests will be run as the Department of Pathology routinely does for all tumor specimens. The normal and cancer tissue left over after the necessary diagnostic tests will be saved in our Tumor Bank and used for the laboratory research measurements related to this study.

One month after your surgical treatment you will meet one more time with your oncologist to have a final physical examination and blood tests to ensure that there is no harm to you from the treatment with durvalumab. After this appointment, no further follow-up for this study will be required.

Testing tissue, both normal and from the tumor, in the lab is one of the main purposes of this study.

You had a biopsy (or surgery) to see if you have cancer. Your doctor has removed a piece of tumor to do tests. The results of these tests were given to you by your doctor and were used to plan your care. At the time of diagnostic biopsy, an extra piece of tumor and neighboring normal tissue might have been removed by your doctor with your consent and deposited in our Tumor Bank. In this case we do not need to repeat the biopsy. If you did not have an extra piece of your tumor removed at the time of first biopsy to be saved in our Tumor Bank, we have to repeat the biopsy after you consent and register with this study. We would like to take an extra piece of your tumor and surrounding normal tissue through a biopsy procedure that is identical with the one that you had initially, at the time of your diagnosis.

Your surgeon will give you local anesthesia. With a syringe and a small needle he will inject a medication to numb you to avoid any pain from biopsy. The medication is the same as you initially had with your first biopsy. Small pieces of tissue will be removed with a punch, scissors or a knife. Sometimes it may be necessary to put in a small, dissolvable suture after the small tumor piece is removed.

The tissue removed through this extra biopsy will be kept and saved in the Tumor Bank in liquid nitrogen and will be used for the research tests approved for this study. Your tumor and normal tissue removed from you by surgical treatment and left over after all the tests carried out by the Department of Pathology for your diagnosis will be also saved in the Tumor Bank and used for the research tests approved for this study

Please read the information sheet called "How is Tissue Used for Research" to learn more about tissue research. This information sheet is available to all at the following web site: <a href="http://www.cancerdiagnosis.nci.nih.gov/specimens/patient.pdf">http://www.cancerdiagnosis.nci.nih.gov/specimens/patient.pdf</a>.

Our nurses can give you a copy at your request.

Your tissue and blood will be used only for research and will not be sold. The research done with your tissue and blood may help to develop new products in the future.

This sample will be kept and may be used in future research to learn more about other diseases.



Your biopsy sample will be obtained in the Hematology and Oncology clinic and your surgical sample will be obtained in the Department of Surgery at Wake Forest University Baptist Medical Center. An Institutional Review Board (IRB) must also approve any future research study using your tissue sample. In order to participate in this study, you must be willing to provide this sample for future research.

Your blood/tissue sample will be stored with a unique identifier and will not include any identifiable information about you such as your name, address, telephone number, social security number, medical record number or any of the identifiers outlined in the HIPAA Privacy Rule. The unique identifier will be a randomly assigned number and only the principal investigator will have access to the code that links the unique identifier to you. Your name, address, social security number, etc., will never be disclosed to future researchers and neither will the code that links your identifiers to the sample.

In the future, people who do research may need to know more about your health. While the study investigator may give reports about your health, he/she will NOT be given your name, address, phone number, or any other identifying information about who you are, unless you agree to be contacted in the future.

| YES you may contact for future research studies | |
|-------------------------------------------------------------------|-----|
| NO I do not want to be contacted regarding future research studie | es. |

#### HOW LONG WILL I BE IN THE STUDY?

You will be in the study for about 90 days after the last dose of Durvalumab.

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences.

## WHAT ARE THE RISKS OF THE STUDY?

#### What is known about the safety of Durvalumab in humans?

Below safety data from 393 subjects with various types of cancer who received Durvalumab alone is provided.

There is a rare risk of presence of blood in bodily fluids: patients can have blood in their sputum (pneumonitis), stool (colitis) or urine (nephritis). Bleeding has been reported in up to 10% or greater in patients with head and neck cancer. Reports of bleeding, including fatal reports, have been received from head and neck cancer patients enrolled in AstraZeneca clinical trials with durvalumab as monotherapy or in combination. It is not yet known whether the risk of bleeding would be higher or lower with the experimental treatment than with standard chemotherapy. Please talk to your study physician immediately if you experience any bleeding. Please also tell your study physician if you are taking any medications that might increase your risk of bleeding, including aspirin, blood thinners, or certain types of pain medications called NSAIDs. Your study physician may suggest that you stop taking these medications while you are on the study drug.



Frequent - Expected to occur in 10% to 25% of people (10 to 25 out of 100 people):

• Fatigue (13.5%)

**Not Frequent** – Expected to occur in 2% to less than 10% of people (2 to less than 10 out of 100 people):

- Nausea (8.4%)
- Diarrhea (5.3%)
- Decreased appetite (5.3%)
- Rash (5.3%)
- Vomiting (4.8%)
- Itchiness (4.1%)
- Difficulty breathing (3.8%)
- Fever (3.1%)
- Low thyroid (2.8%)
- Increased liver enzymes (2.5%)
- Cough (2.5%)
- Muscle pain (2.3%)
- Stomach pain (2.0%)
- Dizziness (2.0%)
- Inflammation of kidney (<1%)
- Inflammation of pancreas (<1%)

**Related** and **serious** side effects reported in subjects receiving Durvalumab alone were:

- Blockage in the urinary tract
- Fluid in the space surrounding the lung and inflammation of the lung
- Increase in calcium in the blood
- Joint pain
- Worsening of cancer
- Increase in liver enzymes and blockage of the tract between the liver and small intestine
- Spinal cord swelling
- Irregular heart beat or rhythm
- Chest pain and fluid in the abdomen
- Dehydration
- Disorder in the blood vessels of the organs
- Swelling of the tumor
- Lack of muscle control during walking or picking up objects
- Inflammation of kidneys with symptoms of blood in urine, low urine output or increased need to urinate, swelling of hands/feet, fatigue)



• Inflammation of the pancreas with symptoms of stomach pain, vomiting, and weakness

The most common long term condition resulting from this treatment is Hypothyroidism, (under active thyroid). The remaining majority of the cases of immunotoxicity heal without long term consequences and respond to steroid treatment.

There was one death felt to be related to Durvalumab when administered alone. The subject who had a prior history of cardiac illness including a prior heart attack died due to a disorder of the blood vessels. The Study Doctor also indicated possible other causes of the fatal event.

A doctor or study nurse will be available to evaluate any side effects and to answer any questions you may have while you are in the study. Clinic staff will be available to answer any questions you may have the day after a dose, and will make arrangements for any evaluations that you might require.

You will be followed closely by your Study Doctor for the entire time you are a part of this study. If you experience one of the side effects listed above or other new side effects, you will be treated right away with the medicines that have the best chance of helping the side effects. If your cancer worsens, you will be treated in the manner you and your Study Doctor feel is best.

If you suffer any of these side effects (or any others not listed) or you think you are experiencing a side effect, during this study, please tell your Study Doctor immediately (see 'Who should you contact for more information?').

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe. In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. There also may be other side effects that we cannot predict. You should tell the research staff about all the medications, vitamins and supplements you take and any medical conditions you have. This may help avoid side effects, interactions and other risks.

For blood draws, you may experience discomfort, bruising and/or bleeding where the needle is inserted. Occasionally some people become dizzy lightheaded or feel faint. Infection may occur on rare occasions. Frequent donation of blood can result in low iron in your blood (iron deficient anemia).

## **Risks Associated With Tissue Biopsy**

Overall the most common risk is bleeding, which can be controlled and stopped in the operating room or clinic.

Infection, a risk of any surgery, is exceedingly rare in the setting of a biopsy.

You can have a reaction to the medication that is used to numb your tumor and the tissue around it, but this is not probable if you did not have any reaction to the first biopsy.



## WHAT DO I HAVE TO DO?

You must be willing to:

- Provide accurate and complete information about your medical history and your present condition.
- Follow the study procedures and keep all scheduled appointments. Inform the study team in advance if you have a problem with keeping an appointment.
- Tell the study team about any other medications (including herbal medications, vaccinations, and over-the-counter medications) you are taking and medical treatments you receive before and during the study. You may not take certain medications or receive certain medical treatments without the permission of the study team during the study or for up to 6 months.
- Tell your Study Doctor about any new side effect, injury, or symptom you experience. Tell
  your Study Doctor of any changes in current medical conditions. This information must be
  reported to your Study Doctor between study visits by using the contact numbers at the end
  of this consent form.
- You should not receive a live vaccination (one that uses live bacteria or viruses) within 30 days before or 30 days after receiving the study drugs.
- If you are female and from the time of informed consent through 1 year following the last dose of study medication you must agree to the following:

# Reproductive Risks and other Issues to Participating in Research

Avoid pregnancy unless you are unable to become pregnant (eg have had your "tubes tied", had a hysterectomy or are at least 1-year post-menopausal). Due to unknown risks and potential harm to the unborn fetus, sexually active women of childbearing potential must agree to use two highly effective methods of birth control as noted in the table below (while taking the study drug and 1 year after that). Reliable methods of birth control are: abstinence (not having sex), oral contraceptives, intrauterine device (IUD), DepoProvera, tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts) in a monogamous relationship (same partner). An acceptable, although less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or a cervical cap or sponge. We encourage you to discuss this issue further with your physicians if you have any questions. Not engaging in sexual activity is an acceptable practice; however, occasional abstinence, the rhythm method and the withdrawal method are not acceptable methods of contraception.

- Refrain from breastfeeding and egg cell donation
- If you are a male subject who is sexually active with a female partner who may become pregnant and from screening through 1 year following the last dose of study medication you must agree to the following:
  - Be unable to get a female partner pregnant (eg. had a vasectomy)
  - If sexually active you must agree to use two highly effective methods of birth control as noted in the table below. Not engaging in sexual activity is an acceptable practice; however, occasional abstinence, the rhythm method and the withdrawal method are not acceptable methods of contraception.
  - Refrain from fathering a child or sperm donation.



• If during the study and through 1 year following the last dose of study medication you learn that you are pregnant (female subject) or your female partner becomes pregnant (male subject), you must contact the Study Doctor immediately for further instructions about follow-up. The study team will ask you about any pregnancy during the study visits and may continue to follow-up with you for up to 180 days after your last dose of study medication. If at any time you report a pregnancy of either you or your partner, the study team will collect information about the results of the pregnancy and/or birth and will schedule any follow-up visits that may be necessary. This health information will become part of the clinical trial records and will be shared with the Sponsor so that the Sponsor may determine if there are any effects of the study medication on unborn children.

#### **Highly Effective Methods of Birth Control**

| | Barrier Methods | Intrauterine device methods | Hormonal Methods |
|---|---|---|---|
| • | Male condom plus spermicide | Copper T | Implants |
| • | Cap plus spermicide | Progesterone T (This is also considered a hormonal method) | Hormone shot or injection |
| • | Diaphragm plus spermicide | | Combined pill |
| | | | Minipill |
| | | Levonorgestrel-releasing intrauterine system (eg, Mirena®) (This also is considered a hormonal method) | Patch |

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. We hope that treatment with Durvalumab might help limit the progression of your cancer until the time of surgery. The information learned from this study will benefit other people in the future.

## WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you can choose to have surgery without treatment with Durvalumab.

## WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you and/or information we get from your medical records about your health or behaviors is considered <u>Protected Health Information</u>. The information we will collect for this research study includes: Demographic information, history of tobacco and alcohol use, medical history, physical exam, performance status assessment, vital signs, height, weight, EKG, current medications, and tumor imaging by CT scan or MRI, PET scan.

If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study will be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with Medical Center operations.



We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer. Only the following people or organizations will be granted access to your Protected Health Information:

- 1) The study investigator and his/her staff, or others at Wake Forest University Health Sciences who oversee research
- 2) Other people or laboratories providing services for this research project on behalf of Wake Forest University Health Sciences and Wake Forest University Baptist Medical Center
- 3) AstraZeneca Pharmaceutical Company, the sponsor of this study.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for an indeterminate period of time. This authorization does not expire. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Dr. Porosnicu that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



Version: 07/11/19 Page **10** of **13** 



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved with this research study.

#### WHAT ARE THE COSTS?

Taking part in this study may lead to added costs to you or your insurance company. We will give you an estimate of what the added cost may be based on your particular situation and insurance coverage. The study drug is provided to you at no cost.

## WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

The purpose of this research study is to obtain data or information on the safety and/or effectiveness of durvalumab; the results will be provided to the sponsor, the Food and Drug Administration and other federal and regulatory agencies as required.



## WILL YOU BE PAID FOR PARTICIPATING?

Parking validation will be provided for all study-related visits.

You will receive no payment or other compensation aside from parking validation for taking part in this study.

The findings from this research may result in the future development of products that are of commercial value. There are no plans to provide you with financial compensation or for you to share in any profits if this should occur.

## WHO IS SPONSORING THIS STUDY?

This study is being sponsored by AstraZeneca Pharmaceutical Company. The sponsor is providing money or other support to Wake Forest University Health Sciences to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

# WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Dr. Mercedes Porosnicu at

## WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study



at any time. This could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions, or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Mercedes Porosnicu at

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at

You will be given a copy of this signed consent form.

#### **SIGNATURES**

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed): | | | |
|-------------------------------------|-------|-------|-------|
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent (Printed): | | | |
| Person Obtaining Consent: | Date: | Time: | am pm |